CLINICAL TRIAL: NCT02243644
Title: A Clinical Trial to Study the Effects of Two Different Duration of Same Drug Albendazole in Patients With Neurocysticercosis in Brain ≤ 5 Lesions on CT Scan Head at the End of 6 Months
Brief Title: Effects of 2 Different Duration of Albendazole Therapy in Patients With Neurocysticercosis in Brain ≤ 5 Lesions on CT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Additional professor, dept of Pediatrics, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IESC/T-320/02.08.2013
Record Dates: First submitted 2014-05-05; First posted 2014-09-18 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Neurocysticercosis
Keywords: parenchymal neurocysticercosis upto five lesions
MeSH Terms: conditions — Neurocysticercosis | interventions — Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): 7 days of albendazole 15 mg/kg/day
  Interventions: Drug: 7 days of albendazole 15 mg/kg/day
- Group B (Active Comparator): 28 days of albendazole 15 mg/kg/day
  Interventions: Drug: 28 days of albendazole 15 mg/kg/day

INTERVENTIONS:
Drug: 7 days of albendazole 15 mg/kg/day — group A will receive 7 days of oral albendazole 15 mg/kg/day
  Other Names: Zentel; Bandy
  Arms: Group A
Drug: 28 days of albendazole 15 mg/kg/day — group B will receive 28 days of oral albendazole 15 mg/kg/day
  Other Names: Zentel; Bandy
  Arms: Group B

SUMMARY:
Comparing the effect of two different duration of same drug albendazole in patients with Neurocysticercosis less than or equal to 5 lesions on CT head at the end of 6 months.

DETAILED DESCRIPTION:
The trial will be comparing the effectiveness of short and long duration of albendazole ie 7 and 28 days therapy in patients with parenchymal neurocysticercosis in terms of complete resolution or calcification of cyst on CT head at the end of 6 months after starting albendazole

ELIGIBILITY:
Inclusion Criteria:

* Age 2-18 years.
* Number of parenchymal lesions: upto 5*
* Stages of cysticerci at which albendazole treatment is effective
* Vesicular stage
* Colloid vesicular stage
* Granular nodular stage

Exclusion Criteria:

* Cysticercotic encephalitis
* Calcified cyst
* Hydrocephalus
* Intraventricular cyst
* Subarachnoid cyst
* Ophthalmic Cysticercosis
* No of cysts >5
* Known allergy to benzimidazole class of compound which includes anaphylaxis, hypotension, severe skin reactions .
* Features of raised ICT (papilloedema, hyperventilation, hypertension, tonic posturing, B/L 6th nerve palsy, features of midline shift on CT/MRI)
* Critically sick (respiratory failure, cardiovascular instability)
* Already received albendazole or praziquantel or steroid therapy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of cyst resolved/ calcified completely after therapy. Resolution or calcification of cyst assessed on CT head at the end of 6 months after starting albendazole | 1 year
  A randomized open labeled control clinical trial to compare the radiological outcome of 7 days versus 28 days albendazole therapy along with steroid in patients with parenchymal neurocysticercosis with lesion load < 5

SECONDARY OUTCOMES:
Frequency of seizure occurrence | 1 year
  A randomized open labeled control clinical trial to compare the radiological outcome of 7 days versus 28 days albendazole therapy along with steroid in patients with parenchymal neurocysticercosis with lesion load < 5
Frequency of occurrence of other symptoms attributable to Neurocysticercosis | 1 year
  A randomized open labeled control clinical trial to compare the radiological outcome of 7 days versus 28 days albendazole therapy along with steroid in patients with parenchymal neurocysticercosis with lesion load < 5
Frequency of occurrence of side effects of albendazole | 1 year
  A randomized open labeled control clinical trial to compare the radiological outcome of 7 days versus 28 days albendazole therapy along with steroid in patients with parenchymal neurocysticercosis with lesion load < 5

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, MD, Principal Investigator — AIIMS, New Delhi
Locations (1):
- sheffali Gulati, New Delhi, National Capital Territory of Delhi, India